CLINICAL TRIAL: NCT06121258
Title: Sexual Health and Breast Cancer: Developing Appropriate Education for Women Going Through Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1734.cc
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female; Sexual Dysfunction
Keywords: Breast cancer; sexual health; educational video
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Video website access (Experimental): Participants will gain access to the educational video website in order to watch the series.
  Interventions: Other: Educational video series

INTERVENTIONS:
Other: Educational video series — The intervention is a web-based educational video series that was developed using a patient-centered approach that discusses breast cancer treatment, sexual health side effects, and provides treatment and mitigation strategies for these side effects.

SUMMARY:
The purpose of this study is to assess the acceptability, appropriateness, and feasibility of a educational video series for patients going through breast cancer treatment.

DETAILED DESCRIPTION:
This is a prospective, mixed methods pilot study to evaluate the acceptability, appropriateness, and feasibility of a novel educational video series for patients going through breast cancer treatment. The video series addresses topics such as what to expect from breast surgery, how to prepare for breast surgery, treatment effects of breast cancer therapies, and mitigation and communication strategies for navigating breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III invasive breast cancer within one month of initial multi-disciplinary clinic visit or surgical consultation
* Ability to complete survey material independently
* Able to read and speak English
* Willingness to comply with study material and procedures

Exclusion Criteria:

* Age < 18 years old
* Stage 0 or IV breast cancer
* Non-breast cancer diagnoses
* History of anti-hormonal therapy, chemotherapy, or radiotherapy not related to breast cancer
* Prior breast cancer diagnosis

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the educational video series after six-months of access and use by breast cancer patients as measured by AIM instrument. | 6 months
  The Acceptability of Intervention Measure (AIM) is a validated instrument used to measure the acceptability of an intervention. Scores range from 0-5. There is no score cut off, however higher scores indicate better outcomes (greater acceptability).
Appropriateness of the educational video series after six-months of access and use by breast cancer patients as measured by IAM instrument. | 6 months
  The Intervention Appropriateness Measure (IAM) is a validated instrument used to measure the appropriateness of an intervention. Scores range from 0-5. There is no score cut off, however higher scores indicate better outcomes (greater appropriateness).
Determine the sustainability of the educational video series after six-months of access and use by breast cancer patients as measured by the FIM instrument. | 6 months
  The Feasibility of Intervention Measure (FIM) is a validated instrument used to measure the feasibility, or sustainability, of an intervention. Scores range from 0-5. There is no score cut off, however higher scores indicate better outcomes (greater feasibility).

SECONDARY OUTCOMES:
Change from baseline in sexual health and function at six-months, as measured by the PROMIS Sexual Function v2 Brief Profile (Female) | Baseline, 6 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sexual Function v2 Brief Profile (Female) is a well-validated tool in oncology patients to assess sexual health. Calibrated subdomain scores are expressed as T-scores (mean=50, standard deviation=10). A T-score 50 corresponds to the mean response among cancer survivors used for previous item testing. Higher scores indicate better outcomes within the domain. We will assess the change at 6 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Tevis, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health, Aurora, Colorado, United States

REFERENCES:
- [Background] Tat S, Doan T, Yoo GJ, Levine EG. Qualitative Exploration of Sexual Health Among Diverse Breast Cancer Survivors. J Cancer Educ. 2018 Apr;33(2):477-484. doi: 10.1007/s13187-016-1090-6. PMID 27492424
- [Background] Sporn NJ, Smith KB, Pirl WF, Lennes IT, Hyland KA, Park ER. Sexual health communication between cancer survivors and providers: how frequently does it occur and which providers are preferred? Psychooncology. 2015 Sep;24(9):1167-73. doi: 10.1002/pon.3736. Epub 2014 Dec 22. PMID 25534170
- [Background] Stead ML, Brown JM, Fallowfield L, Selby P. Lack of communication between healthcare professionals and women with ovarian cancer about sexual issues. Br J Cancer. 2003 Mar 10;88(5):666-71. doi: 10.1038/sj.bjc.6600799. PMID 12618871
- [Background] Stabile C, Goldfarb S, Baser RE, Goldfrank DJ, Abu-Rustum NR, Barakat RR, Dickler MN, Carter J. Sexual health needs and educational intervention preferences for women with cancer. Breast Cancer Res Treat. 2017 Aug;165(1):77-84. doi: 10.1007/s10549-017-4305-6. Epub 2017 May 25. PMID 28547655
- [Background] Huynh V, Vemuru S, Hampanda K, Pettigrew J, Fasano M, Coons HL, Rojas KE, Afghahi A, Ahrendt G, Kim S, Matlock DD, Tevis SE. No One-Size-Fits-All: Sexual Health Education Preferences in Patients with Breast Cancer. Ann Surg Oncol. 2022 Oct;29(10):6238-6251. doi: 10.1245/s10434-022-12126-7. Epub 2022 Aug 1. PMID 35915298
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Flynn KE, Lin L, Cyranowski JM, Reeve BB, Reese JB, Jeffery DD, Smith AW, Porter LS, Dombeck CB, Bruner DW, Keefe FJ, Weinfurt KP. Development of the NIH PROMIS (R) Sexual Function and Satisfaction measures in patients with cancer. J Sex Med. 2013 Feb;10 Suppl 1(0 1):43-52. doi: 10.1111/j.1743-6109.2012.02995.x. PMID 23387911
- [Derived] Higgins MG, Helmkamp L, Zimmaro LA, Leslie SE, Adams M, Vemuru S, Huynh VD, Baurle E, Bozzuto L, Rojas KE, Coons HL, Arkema A, Tevis S. Preliminary evaluation of the acceptability, appropriateness, and feasibility of an online sexual health educational video series for breast cancer patients. Support Care Cancer. 2026 Jan 26;34(2):130. doi: 10.1007/s00520-026-10381-y. PMID 41586882